CLINICAL TRIAL: NCT07153432
Title: Chronic Kidney Disease Screening in Patients Followed at a Tertiary Care Center
Brief Title: Chronic Kidney Disease Screening
Status: Recruiting | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Ondřej Viklický, M.D., Ph.D., Head of Department, Institute for Clinical and Experimental Medicine
Other Study IDs: 23575/25
Record Dates: First submitted 2025-08-06; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; screening; epidemiology
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group
- Control group

SUMMARY:
The goal of this observational study is to assess epidemiology of chronic kidney disease in patients followed at a tertiary care center. The main question it aims to answer is: What is the proportion of patients with chronic kidney disease overall and how many are previously undiagnosed.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 or age >18 + one of these conditions (history of diabetes, arterial hypertension, ischemic heart disease, stroke, perpheral artery disease, atrial fibrillation, heart failure)
* agree to participate
* followed at the Institute for Clinical and Experimental Medicine

Exclusion Criteria:

* unwilling to participate
* kidney transplant recipient/previous kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients followed at the Institute for Clinical and Experimental Medicine
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-10-19 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with chronic kidney disease | Baseline
  Chronic kidney disease diagnosed with either decreased estimated glomerular filtration rate and/or increased albumin excretion in urine

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia